CLINICAL TRIAL: NCT00785265
Title: A Randomized Trial to Reduce the Disparity in Live Donor Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Rodrigue, Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2007P000223; R01DK079665 (NIH)
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Chronic Kidney Disease; End-stage Renal Disease
Keywords: Live Donor Kidney Transplantation; LDKT; African Americans; Disparity; Education
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Based (Experimental): 60-minute group session involving other study patients who have been assigned to this condition and their guests.
  Interventions: Behavioral: Group-Based (GB) Intervention
- Home-Based (Active Comparator): 60-minute educational intervention in their home, which will be delivered by an African American health educator.
  Interventions: Behavioral: Home-Based (HB) Intervention
- Standard Care (No Intervention): 60-minute individual session with an African American health educator.

INTERVENTIONS:
Behavioral: Group-Based (GB) Intervention — 60-minute group session involving other study patients who have been assigned to this condition and their guests.
  Arms: Group Based
Behavioral: Home-Based (HB) Intervention — 60-minute educational intervention in their home, which will be delivered by an African American health educator.
  Arms: Home-Based

SUMMARY:
The main purpose of this study is to learn which educational method is most helpful to patients and their family members when they consider whether to pursue live donor kidney transplantation.

Patients who are eligible for a kidney transplant usually get information in the transplant clinic about two types of kidney transplants - one where the kidney comes from a dead donor and one where the kidney comes from a healthy living donor. Patients are given this information by a transplant nurse or doctor and then encouraged to discuss it with family members and friends.

In this study, we are trying to see if changing how and where we give patients this information makes a difference in how patients and their family members think about live donor kidney transplantation. So, we are looking at whether getting the information in the transplant clinic - either alone or in a group - is the same or different than getting the same information in your home.

The study is only recruiting African American patients. This is being done because African Americans have a higher likelihood of developing chronic kidney disease and needing a kidney transplant than patients of other races. However, they wait longer for a kidney transplant and die at a higher rate on the waiting list because they are less likely than other patients to receive a live donor kidney transplant. We want to see which educational approach works best with African American patients and their families.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) affects over 10 million people in the United States. Diabetes, hypertension, glomerulonephritis, and polycystic kidney disease contribute to most cases of CKD. Those with CKD who become dialysis-dependent are considered to have ESRD. The incidence of ESRD has increased dramatically over the last decade and is estimated to be 338 per million population. Adults with ESRD are known to experience significant mortality and morbidity, and there is evidence of significant health disparities between Whites and ethnic minorities.

While kidney transplantation is the treatment of choice for patients with ESRD, the waiting list and waiting time for deceased donor transplantation are expanding exponentially. Live donor kidney transplantation (LDKT) remains a viable option for patients, yet more than half of all wait-listed patients, especially minorities, do not pursue LDKT. Therefore, programs designed to further expand LDKT, especially those targeting minority populations, are needed given the current and projected shortage of deceased donor organs.

The long-term goal of this research program is to improve education provided to African Americans and, thereby, increase rates of LDKT. The objective of this application is to determine the relative effectiveness of three strategies for increasing LDKT in African Americans. In a recently completed HRSA-funded (2002-2006) randomized clinical trial, we demonstrated that a home-based LDKT intervention program was superior to standard clinic-based education in increasing LDKT rates at one transplant center. The proposed study seeks to replicate and extend the evaluation of a home-based (HB) educational intervention in an African American patient population. The central hypothesis is that a HB intervention yields higher LDKT rates relative to other interventions in African Americans. This hypothesis has been formulated on the basis of strong preliminary data. The rationale for the proposed research is that, by identifying the interventions most likely to yield higher LDKT rates in African Americans, we can further develop and refine the interventional methodology that will allow the most effective education to be disseminated to all kidney transplant programs. We are especially well-prepared to conduct the proposed research due to the multidisciplinary nature of the research team, as well as the expertise and experience of the team in developing LDKT and live donation educational materials, implementing and evaluating novel LDKT interventions, conducting LDKT research with African Americans, and producing meaningful outcomes. Specifically, the research team includes investigators who are funded in the conduct of ESRD, kidney transplantation, and organ donation research and who are dedicated to the scientific advancement of LDKT. Also, the research will be conducted in an environment that is conducive to the successful completion of this project.

To evaluate our central hypothesis and to accomplish the objective of the proposed study, we plan to pursue the following two specific aims:

Specific Aim 1. Determine the clinical effectiveness of three separate LDKT educational approaches with African American patients.

Recently, we found that an LDKT educational intervention delivered in the patient's home and that involved both patients and their invited guests (family, friends, community leaders) was an effective strategy for increasing LDKT, especially in African Americans. This is a very different educational approach than what is used in most transplant centers, which typically involves either group-based (patients and whomever accompanies them to clinic) meetings or individual patient sessions. Based on the work summarized in the Preliminary Studies section, the working hypothesis in this study is that patients randomized to a Home-Based (HB) intervention will demonstrate more favorable outcomes relative to patients randomized to a Group-Based (GB) intervention conducted in the transplant clinic or to a Standard Care (SC) condition in which individual patients are education in the transplant clinic. Specifically, relative to the GB or SC educational approaches, the HB intervention will demonstrate...

Primary Outcome:

Hypothesis 1.1: A higher proportion of enrolled patients with LDKTs.

Secondary Outcomes:

Hypothesis 1.2: A higher proportion of enrolled patients with live donor inquiries.

Hypothesis 1.3: A higher proportion of enrolled patients with live donor evaluations.

Hypothesis 1.4: A higher number of potential donors educated, per patient. Hypothesis 1.5: More improvement in live donation knowledge. Hypothesis 1.6: More improvement in live donation concerns. Hypothesis 1.7: More willingness to initiate live donor discussion with others.

Specific Aim 2. Determine the sociodemographic, medical, and donation-specific variables that are most strongly associated with pursuing LDKT.

Based on the work summarized in the Preliminary Studies section, the working hypothesis is that LDKT status (primary outcome: yes/no) will vary significantly by sociodemographic, medical, and donation-specific variables. Specifically… Hypothesis 2.1: The following patient characteristics will be significantly associated with having received LDKT: male, younger, dialysis-dependent, more live donor inquiries, more knowledge about live donation, fewer concerns about live donation, and more willingness to initiate live donation discussion with others.

ELIGIBILITY:
Inclusion Criteria:

* African American race
* male or female
* 21 to 80 years old
* diagnosis of ESRD
* eligible for listing on the kidney transplant waiting list at Beth Israel Deaconess Medical Center
* resides within 150 minutes of transplant center
* residential or cell phone service
* signed informed consent

Exclusion Criteria:

* Wait-listed for additional organ transplant (i.e., heart, liver)
* current substance abuse or dependency
* known or suspected psychotic disorder
* known or suspected mental retardation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2007-08; Primary Completion 2015-11 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome for this study is the proportion of enrolled patients with live donor kidney transplants. | one year

SECONDARY OUTCOMES:
Higher proportion of enrolled patients with live donor inquiries and evaluations; and higher number of potential donors educated. Improvement in live donation knowledge, concerns, and willingness to initiate live donor discussion with others. | one year

CONTACTS AND LOCATIONS:
Overall Officials: James R Rodrigue, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center; Martha Pavlakis, MD, Study Chair — Beth Israel Deaconess Medical Center; Didier Mandelbrot, MD, Study Chair — Beth Israel Deaconess Medical Center; Ogo Egbuna, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- [Derived] Rodrigue JR, Pavlakis M, Egbuna O, Paek M, Waterman AD, Mandelbrot DA. The "House Calls" trial: a randomized controlled trial to reduce racial disparities in live donor kidney transplantation: rationale and design. Contemp Clin Trials. 2012 Jul;33(4):811-8. doi: 10.1016/j.cct.2012.03.015. Epub 2012 Apr 3. PMID 22510472